CLINICAL TRIAL: NCT06038409
Title: Understanding the Safety of Home Ketamine Treatment Plans for Chronic Conditions
Brief Title: Ketamine Treatment Plans for Chronic Conditions
Status: Recruiting | Type: Observational
Sponsor: RIVER Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: RIVERFoundation 001
Record Dates: First submitted 2023-01-01; First posted 2023-09-14 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-01

CONDITIONS: Chronic Pain; Depressive Disorder; Anxiety Disorders; Chronic Disease
MeSH Terms: conditions — Chronic Pain; Depressive Disorder; Anxiety Disorders; Chronic Disease | interventions — Ketamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Chronic Pain: The use of ketamine in chronic pain
  Interventions: Drug: Ketamine
- Depressive Disorders: The use of ketamine in depressive disorders
  Interventions: Drug: Ketamine
- Anxiety Disorders: The use of ketamine in anxiety disorders
  Interventions: Drug: Ketamine
- Chronic Condtions: The use of ketamine in chronic conditions
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — The efficacy of the various approaches to prescribing Ketamine currently in use off-label. The focus will be to include ketamine within the treatment plan of those with chronic conditions

SUMMARY:
A study aimed to assess the efficacy of the various approaches to prescribing Ketamine currently in use off-label. The focus will be to include ketamine within the study plan of those with chronic conditions who are receiving ketamine.

DETAILED DESCRIPTION:
Ketamine can be administered in multiple ways (IV, IM, SubQ, and Sublingual, among others), and there have been few if any, studies that have compared the impact of Ketamine at home without any thearpy.

The study will identify other treatment modalities used in concurrence with Ketamine. Psychotherapy, music therapy, and acutherapy are some of the most popular. How do these adjunct therapies affect the outcomes of Ketamine treatments?

Secondarily, the study will focus on these significant issues to observe the impact of Ketamine treatments and suicidal ideation. Suicidal ideation is multifaceted and is one reason for prescribing off-label Ketamine. Chronic issues such as depression, pain, and anxiety have been identified as underlying causes and may be improvable with Ketamine.

ELIGIBILITY:
Inclusion Criteria:

Must have an identifiable chronic condition.

Exclusion Criteria:

Healthy population

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with chronic conditions that need either their mental health or pain controlled.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Ketamine route of use acceptability. | through study completion, an average of 1 year
  Compare and Contrast the different methods and uses of ketamine for acceptability for the route of use. (ie oral sublingual or nasal spray)
Mental Health PHQ9 | through study completion, an average of 1 year
  The use of psychological scales to measure participants' mental health with the use of ketamine. Three scales will be charted to examine the mental health of the participant.
  The Patient Health Questionnaire-9 (PHQ9), Patient Health Questionnaire 9 has a possible range of 0-27. Zero being no depression and 27 being severe depression.
  Participants will be given a baseline survey and will be given a survey to complete every time they request a ketamine renewal while participating in the study. A multiline graph will show the results of the amount of ketamine and the PHQ9 will be produced.
Mental Health GAD7 | through study completion, an average of 1 year
  Participants will be screened using the Generalized Anxiety Disorder-7 (GAD7) with a total score for the seven items ranging from 0 to 21. Scores 5, 10, and 15 represent cut points for mild, moderate, and severe anxiety, respectively.
  Participants will be given a baseline survey and will be given a survey to complete every time they request a ketamine renewal while participating in the study. A multiline graph will show the results of the amount of ketamine and the GAD7 will be produced.
Mental Health PCL5 | through study completion, an average of 1 year
  Participants will be screened using the Posttraumatic Stress Disorder Checklist (PCL-5) PCL-5. On a 4-point scale, scores can be tabulated for individual items to give information about the severity of the four DSM-5 symptom clusters. If a score of 2 (moderate) is considered to be a positive endorsement of a given criterion, the PCL-5 can be used in combination with a clinical interview to make a provisional DSM-5 diagnosis. Testing the PCL-5 with veterans has determined a score of 31 to 33 to be a valid cutoff for a positive screen. The scores range from 0-80, 0 being no symptoms to extreme issues with post-traumatic stress disorder.
  Participants will be given a baseline survey and will be given a survey to complete every time they request a ketamine renewal while participating in the study. A multiline graph will show the results of the amount of ketamine and the PCL5 will be produced.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Lesofski, MS, Study Director — RIVER Foundation
Locations (1):
- RIVER Telehealth, Helena, Montana, United States

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- See also: RIVER's research web site — http://research.riverofchange.org